CLINICAL TRIAL: NCT04777006
Title: Integrating a Stepped Care Model of Screening and Treatment for Depression Into Malawi's National HIV Care Delivery Platform
Acronym: IC3D
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Partners in Health (Other); Brigham and Women's Hospital (Other); Malawi Ministry of Health (Unknown); Blantyre College of Medicine (Unknown); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH117760 (NIH)
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder
Keywords: depression; stepped care; behavioral therapy; Problem Management Plus; antidepressant therapy
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Fluoxetine; Amitriptyline

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Those who are screening and diagnosing depression will not be made aware of the randomization sequence. Likewise, those assessing outcomes will not be made aware of the randomization sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cluster 1 (First Cluster of Clinics Randomized to Receive Care) (Experimental): Arm 1 represents a cluster of 2-3 clinics randomized to begin delivering the intervention at month 3 of the trial
  Interventions: Behavioral: Problem Management Plus; Drug: Antidepressant Therapy
- Cluster 2 (Second Cluster of Clinics Randomized to Receive Care) (Experimental): Arm 2 represents a cluster of 2-3 clinics randomized to begin delivering the intervention at month 6 of the trial
  Interventions: Behavioral: Problem Management Plus; Drug: Antidepressant Therapy
- Cluster 3 (Third Cluster of Clinics Randomized to Receive Care) (Experimental): Arm 3 represents a cluster of 2-3 clinics randomized to begin delivering the intervention at month 9 of the trial
  Interventions: Behavioral: Problem Management Plus; Drug: Antidepressant Therapy
- Cluster 4 (Fourth Cluster of Clinics Randomized to Receive Care) (Experimental): Arm 4 represents a cluster of 2-3 clinics randomized to begin delivering the intervention at month 12 of the trial
  Interventions: Behavioral: Problem Management Plus; Drug: Antidepressant Therapy
- Cluster 5 (Fifth Cluster of Clinics Randomized to Receive Care) (Experimental): Arm 5 represents a cluster of 2-3 clinics randomized to begin delivering the intervention at month 15 of the trial
  Interventions: Behavioral: Problem Management Plus; Drug: Antidepressant Therapy

INTERVENTIONS:
Behavioral: Problem Management Plus — PM+ is a cognitive-behavioral intervention that trains recipients to improve their management of practical problems, and uses the term "problem management" rather than "problem solving" to emphasize that many problems encountered by individuals living in adverse circumstances may not be "solvable". The "plus" in PM+ underscores additional evidence-based behavioral strategies incorporated into the model, including: stress management strategies, behavioral activation, and social support strengthening. In total, PM+ comprises five sessions held once per week for 1.5. to 2.5 hours per session. The model has shown success in reducing depression symptoms in low-resource settings such as Nepal and Pakistan.4
  Other Names: PM+
Drug: Antidepressant Therapy — Fluoxetine, a serotonin selective reuptake inhibitor (SSRI), and amitriptyline, a tricyclic antidepressant (TCA), are part of Malawi's national formulary. Neno District supply chain is supported by PIH, which reduces stock-outs relative to those observed in other Malawian settings. Fluoxetine is typically the first drug of choice because it is safer and better tolerated.
  Daily dose will commence at 20 mg of fluoxetine, or 25 mg of amitriptyline. At monthly follow-up visits, a dose increment or medication change may be considered based on measures of treatment response and side effects, using an Antidepressant Side Effect Checklist. This algorithm-based process will be repeated every other week until the patient is fully responding to treatment (PHQ-9 < 5) for a period of three months. Dose escalations of more than one increment and medication changes will be reviewed with the doctor-in-charge. If on ADT at end of study, it will be sustained as part of usual care.
  Other Names: Fluoxetine; Amitriptyline

SUMMARY:
Malawi is a low-income country in sub-Saharan Africa that has limited resources to address a significant burden of disease-including HIV/AIDS. Additionally, depression is a leading cause of disability in the country but largely remains undiagnosed and untreated. Lack of cost-effective, scalable solutions is a fundamental barrier to expanding depression treatment. Against this backdrop, one major success has been the scale-up of a network of more than 700 HIV clinics, with over half a million patients enrolled in ART. As a chronic care system with dedicated human resources and infrastructure, this presents a strategic platform for integrating depression care, and responds to a robust evidence base outlining the bi-directionality of depression and HIV outcomes.

The investigators will evaluate a stepped model of depression care that combines group-based Problem Management Plus (group PM+) with antidepressant therapy (ADT) for 420 adults with moderate/severe depression in Neno District, Malawi, as measured by the Patient Health Questionnaire-9 (PHQ-9). Rollout will follow a stepped-wedge cluster randomized design in which 14 health facilities are randomized to implement the model in five steps over a 15-month period. Primary outcomes (depression symptoms, functional impairment, and overall health) and secondary outcomes (e.g. HIV: viral load, ART adherence; diabetes: A1C levels, treatment adherence; hypertension: systolic blood pressure, treatment adherence) will be measured every three months through 12-month follow-up. The investigators will also evaluate the model's cost-effectiveness, quantified as an incremental cost-effectiveness ratio (ICER) compared to baseline chronic care services in the absence of the intervention model.

This study will conduct a stepped-wedge cluster randomized trial to compare the effects of an evidence-based depression care model versus usual care on depression symptom remediation as well as physical health outcomes for chronic care conditions. The investigators will also look at the indirect effects of the intervention at the household level. The investigators' hypothesis is that the intervention will be effective at reducing depression symptoms, improving physical health, and improving household members' wellbeing, compare to treatment as usual. The investigators also hypothesize that the intervention will be highly cost-effective, meaning that the cost per QALY gained will be less than Malawi's median GDP per capita. If determined to be effective and cost-effective, this study will provide a model for integrating depression care into HIV clinics in additional districts of Malawi and other low-resource settings with high HIV prevalence.

DETAILED DESCRIPTION:
BACKGROUND

Major depressive disorder imposes catastrophic health and economic impacts in Malawi, and throughout sub-Saharan Africa. Depression is a leading cause of disability in Malawi. Yet, best evidence suggests that over 90% of individuals with the condition receive no treatment (1). The cost of inaction is liable to have wide-ranging impacts. In terms of health, depression-when untreated-typically observes a recurrent trajectory across the lifespan, and is associated with significant depreciation in quality of life. Depression also indirectly impacts other health outcomes, including HIV outcomes such as adherence to antiretroviral therapy and health-seeking behavior. In terms of social ecology, depression affects interpersonal relationships, engagement in household activities, and labor force participation. The World Economic Forum has estimated a $30 trillion loss over a twenty-year span due to neglected treatment of neuropsychiatric conditions, largely due to lost labor force participation (2).

Integrating depression care into Neno's HIV platform represents a cost-effective, scalable solution in Neno District, Malawi, consistent with best practices. Over the past 10 years, Malawi has enrolled over a million individuals in antiretroviral therapy. Current enrollment levels stand at 580,000. This has been achieved by introducing a framework of HIV care delivery, the basis of which is a network of 706 HIV clinics throughout the country. Over this same timeframe, HIV has evolved from an acute condition with poor prognosis, to a chronic condition with vastly improved survival rates. Given this context, the HIV system is a strategic point of entry for screening and treating depression, as it represents a leveragable chronic care system. In Neno District, HIV facilities have already transitioned into an integrated chronic care platform for treating conditions like diabetes, hypertension, asthma and epilepsy. Likewise, community health screenings, routine in Malawi, could be leveraged to screen for depression.

Overarching Objective. Evaluate a clinical model of screening and treatment for depression in terms of 'real world' effectiveness and cost-effectiveness at reducing depression in Neno District.

Objective 1. Determine the implementation strategy effectiveness-in terms of improved depression (PHQ-9), daily functioning (WHODAS), and overall health (EQ5D)-of introducing a stepped model of depression care (behavioral therapy and antidepressant therapy) among adults receiving integrated chronic care in Neno District, Malawi between July 1, 2021-June 30, 2025.

Objective 2. Determine the cost-effectiveness the stepped model of depression care (behavioral therapy and antidepressant therapy) among adults receiving integrated chronic care in Neno District, Malawi between July 1, 2021-June 30, 2025.

Objective 3: Assess positive externalities associated with depression care, including improved wellbeing among household members of treated patients, and improved physical health outcomes among patients receiving depression care.

Objective 4: Inspect mediators and moderators of improved depression care, including a dose effect from level of treatment received (number of behavioral therapy sessions), reduced internalized mental health stigma, and improved perceived social support.

RATIONALE

The framework strategically addresses the bi-directionality of depression and HIV outcomes. A broad literature throughout sub-Saharan Africa has outlined the impact of HIV-including HIV-related stigma, reduced quality of life and ability to maintain employment-on elevated depression levels (3). Depression, in turn, predicts HIV-related outcomes such as adherence to ART. As such, targeting depression care among a population that includes HIV+ individuals in Malawi should yield significant benefits in terms of HIV-related outcomes. Outside sub-Saharan Africa, there is increasing evidence that integrative health services represents stronger value for money than stand-alone models.

Research examining the benefits and costs of treating neuropsychiatric conditions, including depression, suffers two key limitations. First, evaluations have only measured individual-level, direct treatment effects. This approach under-appreciates the social ecology of mental health: that individuals are typically situated within families, and families within communities. From this lens, neuropsychiatric disorders have shown adverse effects-in terms of burden of care and emotional wellbeing-on household members. Previously, the investigators showed that, when individuals' mental health improves through treatment, indirect benefits are observed among household members (4). Likewise, measurement limited to direct treatment effects overlooks indirect benefits to overall health, including for comorbid conditions such as HIV, that may result from mental health intervention. A second shortcoming is that evaluations have focused on measuring costs of standalone interventions, which are costlier than those that leverage existing systems. For instance, interventions for youth have often integrated within school systems to lower costs. In Malawi, the national HIV system-already transitioning to an integrated chronic care platform in Neno District-holds potential to treat depression at lower costs by building on established systems of longitudinal care.

In terms of historical objectives, a preponderance of mental health evaluations in low-resource settings has stopped at the point of measuring effectiveness, rather than cost-effectiveness, with a few exceptions by project members. The consequences are marked: In settings of financial constraint such as Neno District, Malawi, resources allocated to a particular program necessarily means resources allocated away from another. As such, assessing intervention costs are fundamental for determining scalability. A collaborative care model of treatment for depression and comorbid conditions such as HIV and diabetes has the potential to overcome resource constraints, which cost-effectiveness analysis would demonstrate.

The investigators will evaluate an evidence-based stepped care model of depression treatment integrated into Neno's HIV system, assessing health outcomes and cost-effectiveness, inclusive of direct and indirect benefits. Partners In Health (PIH), in collaboration with the Malawian Ministry of Health, has operated in Neno District-home to 165,000 Malawians-for 12 years. The investigators proposed to integrate a stepped care model for depression-combining antidepressant therapy (ADT) with group-based Problem Management Plus (PM+), the elements of which have been successfully instituted by the research team in low-resource settings, ranging from Rwanda to Haiti. The proposed study will evaluate a model that trains clinical staff situated in clinics to screen and diagnose depression, and administer PM+ among those with a diagnosis of moderate or severe depression. Over five weekly 1.5-2.5 hour group sessions, the behavioral intervention combines empirically-based treatment components such as psychoeducation, strategic problem solving, and behavioral activation (5). This will be coupled with antidepressant therapy (ADT) among those with severe depression.

To assess intervention benefits, the investigators will measure patient outcomes for depression every 3 months-including baseline, post-intervention, 6-months, and 12-months follow-up-as well as markers of comorbid conditions: including viral load and ART adherence among those are HIV+ (71% of the sample) as well as other disease-specific outcomes such as systolic blood pressure for hypertensive patients (17% of sample) and hemoglobin A1C for diabetic patients (2% of sample)-supported by an electronic medical records system. Importantly, to quantify indirect benefits of depression care, the investigators will also interview household members at baseline and 6-months follow-up to evaluate burden of care, including emotional distress and missed days of work. The investigators will convert direct and indirect benefits to quality-adjusted life years (QALYs).

METHODS

Design of Study. We will implement a stepped-wedge cluster randomized trial of an evidence-based intervention for depression care within Neno's HIV system, currently undergoing transition to a chronic care platform, examining depression symptoms and outcomes of comorbid conditions, inclusive of HIV, across 14 facilities rolled-out clinic-wide in five steps over 15 months (6). This design is a gold standard experimental approach aligned with PIH's clinical goal to implement depression care permanently throughout Neno District, and is a methodological framework on which we have unique expertise, including locally.

Place of Study. This study will take place in Neno District, a catchment area of 165,000 Malawians, where 12,186 are enrolled in integrated chronic care-including for HIV. Five-year retention in ART in Neno District is 80%, while five-year mortality is close to 15%. The viral suppression rate is 83%. These figures signify Neno as high performing but also underscores significant room for improvement-particularly among the most vulnerable, such as those with depression. As such, we do not anticipate a ceiling effect for measuring HIV outcomes among those concurrently enrolled in depression care. This is also true for other chronic conditions: e.g. only 60% of hypertensive patients currently have controlled systolic blood pressure (<140 mm Hg). Successes to-date have been achieved through modest human resource investments such as CHWs, suggesting replicability nationally. This has been supported by the investigators' past cost-effectiveness analyses.

Target Population. The investigators intend to recruit at least 420 adults with depression for participation in this study, beginning July 1, 2021 and continuing through June 30, 2025. This number is based on the sample size needed for us to determine the effectiveness of the depression treatment, as well as the prevalence of depression in Malawi: At each ICC clinic, 200-1,800 patients are seen on a quarterly basis. The investigators anticipate 10%-12% of all patients (n=12,186) will screen positive for depressive symptoms, and 6% will be diagnosed with moderate/severe depression. Prior studies in Malawi have found acceptance of research study participation is 90% or higher. In addition, the investigators will be conducting interviews with 210 households among half of participants-in order to determine whether the intervention improves quality of life within households.

Sampling Techniques and Tools. The full study period is January 1, 2021 through June 30, 2025. The first six months will be preparation. Beginning July 1, 2021, all adults attending integrated chronic care clinics will be screened for depression symptoms using the PHQ-2 by existing clinical officers. Consistent with the prior screening literature, those with a score > 2 will complete remaining questions of the PHQ-9; and a score >9 will trigger administration of a brief diagnostic interview--adapted from the CIDI 3.0--by a trained counselor. Those with PHQ-9<10 (no/mild depression) will receive a psychoeducation session, but will not be enrolled-based on limited availability of health professionals and need-based prioritization. Those with moderate/severe depression (PHQ-9>9, corresponding to diagnosis of major depression) will be eligible for cohort enrollment. Screening, diagnosis and enrollment will occur continuously across all facilities over the full trial period; those who meet diagnostic criteria will be enrolled. Treatment will be rolled-out progressively: patients in each cluster's cohort will be initiated into the intervention: Three facilities will begin treatment immediately (Step 1), with remaining facilities will initiate treatment at three- (Step 2), six- (Step 3), nine- (Step 4) or twelve-months (Step 5) later. The stepped-wedge approach enables all facilities throughout Neno District to implement the model, as such maintaining equipoise. Assessment of patients on outcome measures will occur at every 3 months.

Sample Size Determination. The investigators assume n=30 enrollees per facility (total n=420), based on depression prevalence in Malawi. The investigators further assume loss to follow-up of 15%, based on intervention trials that the investigators have conducted in similar settings. To account for clustering, the investigators calculated detectable differences using an intracluster correlation coefficient (ICC) of 0.05 within treatment group and 0.01 within rollout step, based on depression treatment studies in multiple developing countries, including the investigators' pilot work. Based on this, the investigators find n=420 enrollees to be sufficient (power > 0.80; (alpha=.05; 2-tailed) for detecting a clinically meaningful standardized effect size of 0.5 (Cohen's d) for primary outcomes, including accounting for cluster autocorrelation. This is not separated by modality (though the investigators will explore this): it is to assess overall effectiveness of the stepped care model.

Data Collection Techniques and Tools. Over the 15-month roll-out period, primary outcomes (PHQ-9, WHODAS, EQ5D) will be measured at three-month intervals among all participants from point of enrollment, consistent with the three-month increments between steps (see above). Three-month increments will coincide with treatment initiation, post-intervention, 6 months and 12 months follow-up. In the event an enrolled individual no longer meets criteria at treatment initiation, the individual will leave the cohort and not be eligible for treatment but will continue to be evaluated every three months for future eligibility. Given that screening, diagnosis and enrollment will occur at all facilities over the full trial period, the investigators expect any reduction in patients enrolled in the cohort due to lagged treatment initiation will be offset by newly-identified individuals over this same period. This is consistent with an open cohort design for stepped-wedge trials. Ultimately, this approach enables all facilities to implement the model, maintain equipoise, and create control sites by randomizing roll-out sequence. Measurement intervals are consistent with best practices in outcomes tracking, including past trials. Interviews with household members will be conducted at treatment initiation and 6-month follow-up, among 210 randomized households.

Data Analysis. Analysis will assume a mixed-effects longitudinal regression framework, which the team has implemented in similar contexts. To account for nesting of patients within treatment groups and clusters, as well as time points (autocorrelation), patient, patient group and cluster will be incorporated as random effects, while cluster assignment and covariates are included as fixed effects-using STATA's MIXED command. The investigators will run sensitivity analyses to test if data are missing at random (MAR), and examine stigma and social support as moderators, as well as potential mediation using causal mediation analysis.

Effectiveness. The investigators will use linear mixed-effects regression analysis to test differences between study arms on change in primary outcomes. Models will adjust for patient demographics, as well as stigma and social support. Analysis will assume an intention-to- treat (ITT) framework, with and without multiple imputation analysis. In addition to ITT, the investigators will perform a 'completers only' analysis to exam outcomes among those who adhered to treatment, and examine dose response.

Cost-effectiveness. Health measures will be converted to QALYs using the EQ5D-3L cross-walk between domain-specific outcomes. This approach has been utilized and published on previously. QALY estimates will be related to base case and treatment cost estimates. For formal CEA, the investigators will use a gold standard Markov chain Monte Carlo (MCMC) simulation-based approach in TreeAge, from a societal perspective. For sensitivity analyses, the investigators will vary discount rates from 0-5%, based on health-adjusted life expectancy. Unit of interest is the incremental cost-effectiveness ratio (ICER) of cost per QALY, comparing the cost of integrated chronic care before and after introduction of the depression treatment.

PROTOCOL

Evidence-based treatment of depression. Drawing from a manual-driven framework of enhanced Problem Solving Therapy (PST) known as Problem Management Plus (PM+), developed by the WHO for low-resource settings, the investigators will implement a gold standard, stepped approach to treatment for depression. The model will follow a group format, based on three considerations: this lowers costs of human resources, which is essential when considering national scalability; it provides peer support during treatment; and it is culturally appropriate for the setting. These considerations have been sources of advocacy for the group model by WHO. In settings where group format has been implemented, results have been comparable to individual format. Local counselors will administer PST in five 1.5-2.5 hour sessions, with 6-8 participants per group, consistent with WHO guidelines. Among those with PHQ-9>15, antidepressant therapy (ADT) will be offered following WHO mhGAP procedures.

Depression screening. The investigators will screen patients ages 18+ enrolled in ICC clinics in Neno District, beginning the first quarter of Y2. Screening, diagnosis and enrollment into the treatment cohort will occur continuously across facilities, administered by data clerks and counsellors trained on the PHQ-2 and PHQ-9, respectively (6). Screening will also occur every 3 months among individuals in the active cohort to determine current treatment eligibility status. The PHQ-2 assesses frequency of depressed mood and anhedonia, and has been implemented throughout Africa. Use of PHQ-2 as a first step has will save time: the investigators are screening 12,186 adults. The selected threshold allows high sensitivity. Patients who screen positive with the PHQ-2 (score >2; range: 0-6) will immediately receive remaining PHQ-9 questions, on which a score > 9 (range: 0-27) represents a possible depressive disorder. Those with PHQ-9<10 will receive a psychoeducation session from the clinical officer, using a manual on which they have been trained. Those with PHQ>9 (moderate/severe depression) will be referred to a counselor to administer the diagnostic protocol.

Depression diagnosis. Counselors will review PHQ-9 scores and administer a brief diagnostic interview--based on the Comprehensive International Diagnostic Interview (CIDI)--to diagnose depression: 5 of 9 symptoms present and functional impairment. All patients will be evaluated for suicide risk and whether immediate intervention is warranted. If so, they will be referred to the supervising physician at the health facility, triggering an emergency protocol. Patients will be assigned to one of three categories: mild, moderate and severe depression. Those with a negative diagnosis will not be eligible for the intervention, and will undergo PHQ-2 screenings at subsequent visits for eligibility. Those with a positive diagnosis and PHQ-9>10 will be eligible. Those with PHQ-9 10-14 will be offered PST alone. Those with PHQ-9>15 (moderate-to-severe depression) will be offered PST and ADT as joint treatment, with the alternative to choose a single modality. Pregnant women with severe depression will also be eligible for ADT. Best evidence, including recent systematic reviews, does not find increased risk for mother or infant with appropriately administered ADT, and there are significant potential benefits of improved wellbeing of the mother.

Psychoeducation and treatment selection. Counselors will inform patients on availability of PST and ADT, outline potential benefits and risks, provide an overview of the study, and acquire informed consent. Those who decline care will be offered psychoeducation and referred to available resources. Among those who elect PM+, the first PM+ session will also incorporate in-depth psychoeducation. Patients with a PHQ-9 score of 10-14 will be provided the option of ADT but recommended PM+ instead, given that behavioral therapy has established efficacy and avoids potential side effects of ADT. Patients with PHQ-9 > 15 will also be given the options of PST, ADT, or both, and recommended both. At facilities randomized to administer the intervention immediately, patients will be informed of date, time and location of their first PM+ session.

Problem Management Plus (PM+). Counselors (n=8) will receive intensive training in Year 1 by to administer PM+ using a manualized approach. Training and supervision are described below. PM+ is a WHO-enhanced framework of Problem Solving Therapy (PST) for implementation by lay personnel in low-resource settings like Neno, designed to be conducted in five weekly 1.5-2.5 hour sessions. Elements of PM+, including sequential problem solving, have been applied by the research team in numerous settings with marked success, including in Lilongwe. This district-wide randomized trial leveraging Neno's existing infrastructure would represent a critical evidential support for WHO's agenda to expand the model globally. Modules include: psychoeducation, managing problems, behavioral activation, social support strengthening, and stress reduction.

Antidepressant Therapy (ADT). The investigators expect 20-25% of study participants-i.e. those who meet diagnostic criteria-to have moderately severe or severe depression and opt to enroll in ADT. Fluoxetine, a serotonin selective reuptake inhibitor (SSRI), and amitriptyline, a tricyclic antidepressant (TCA), are part of Malawi's national formulary. Neno District has a robust supply chain, which will reduce stock-out. Potential side effects of ADT are modest but include nausea, insomnia, and nervousness and will be communicated to participants prior to initiation. There is modest evidence ADT may increase risk of suicidality; this risk will be stated in informed consents, counselors will be trained to identify this risk, and will be formally assessed during outcome assessments, with the potential to trigger protocol for suicidal ideation. Benefits of ADT often outweigh risk of harm and negative impact of untreated depression. Fluoxetine is typically the first drug of choice because it is better tolerated.

Dosing Algorithm: Daily dose will commence at 20 mg of fluoxetine, or 25 mg of amitriptyline. Dose increments and levels are the same for each drug. At monthly follow-up visits, a dose increment or medication change may be considered based on measures of treatment response and side effects, using the Antidepressant Side Effect Checklist. This algorithm-based process will be repeated bi-weekly until the patient is fully responding to treatment for a period of three months (PHQ-9 < 5). Dose escalations of more than one increment and medication changes will be reviewed with the doctor-in-charge.

MEASUREMENT

Primary Outcomes. Measures will include surveys, laboratory assays, pharmacy data, and data abstracted from medical charts and the Depression Care Registry. Survey measures that have not been translated into Chichewa in the course of prior research will be translated using standard translation, back-translation methods, and will be administered at each assessment, unless otherwise noted.

Depression symptoms. Depression symptoms will be measured with the PHQ-9, which has been translated previously and locally-validated. The investigators have elected to use PHQ-9 because it has been implemented throughout sub-Saharan Africa, including Malawi, where the scale has shown high sensitivity responding to treatment, as well as concurrent and predictive validity. It contains nine four-point ordinal response items on topics such as hopelessness, psychosomatic response (e.g. sleeplessness, loss of appetite) and anhedonia.

Functional impairment. Functional impairment including aspects of daily functioning, correspond to DSM diagnostic criteria. The investigators will evaluate this using the 12-item WHO Disability Assessment Schedule 2.0 (WHODAS). The WHODAS has been validated in a diverse range of sub-Saharan African contexts, including Malawi, and covers topics like completing household chores, concentrating, and maintaining relationships.

Overall health. A health profile will be generated for each individual using the EQ-5D-3L, previously validated in Malawi. This survey determines patients' overall health at time of interview and offers a cross-walk to quality-adjusted life years (QALYs).

Secondary Outcomes. Secondary outcomes will constitute those measuring indirect benefits and costs of treatment. Indirect benefits will be incorporated into cost-effectiveness estimates by internalizing improvements among comorbid conditions such as HIV and hypertension, as well as reduced household burden of care.

ART adherence. ART adherence will be measured in terms of whether HIV+ enrollees have returned to an IC3 for antiretrovirals (ARVs) within the past three months, an approach considered more reliable than self-reports. This interval overlays with clinical protocols throughout Malawi in terms of the duration for which ARVs are supplied.

Viral load. Viral load will be measured as part of HIV+ patients' clinical assessment pre-intervention, post-intervention, 6- and 12-month follow-up, consistent with ongoing care at IC3s. This is considered a key metric for determining treatment plans and is highly sensitive to compliance with prescribed ART regimens.

HIV disease staging. Staging will be evaluated every three months among HIV+ enrollees, consistent with IC3 visits. This approach to tracking disease progression is commonly used in low-resource settings.

Chronic care outcomes. Chronic care outcomes on hypertension, type-2 diabetes, and epilepsy will be abstracted from electronic medical records. Systolic blood pressure and adherence to antihypertensive medication (measured by medicine pickups) will be measured among those with hypertension. Among those with type-2 diabetes, adherence to quarterly visits and A1C (or random blood sugar) levels will be abstracted. Among those with epilepsy, the investigators will catalog number of reported seizures in past quarter, and adherence to antiepileptics as measured by quarterly medicine pickups.

Household burden of care. Lastly, household burden of care will be evaluated with household members using a locally-adapted version of the Burden Assessment Schedule (BAS), previously implemented by the team. The survey assesses dimensions of emotional and functional burden of care, including missed work, guilt and worry.

Mediators and Moderators. Analyses will also include three mediators/moderators assessing potential pathways by which depression treatment leads to alleviation of depression symptoms, including enhanced social support, reduced HIV and depression-related stigma, and performance of psychosocial counsellors as quantified by fidelity to PM+ protocols.

Perceived social support. Social support strengthening is a focus of PM+. This will be measured with the Multidimensional Scale of Perceived Social Support (MSPSS), previously validated, to assess support before and after care.

Perceived stigma. Self-perceived stigma is associated with HIV status and depression, including in Malawi. The investigators will adapt the AIDS-Related Stigma Scale (ARSS) and Internalizing Stigma of Mental Illness (ISMI) scale in Year 1 of the project-both designed for use in community-based settings in sub-Saharan Africa.

PM+ fidelity. Fidelity checklist scores will be generated for each counsellor by a lead clinical officer or supervisor. Research has shown that fidelity protocols are predictive of patient outcomes in the context of depression care.

Household Interviews. Adult household members of participants-one per household-will be identified for participation based referral by the study participant and/or self-identification as a social support in close contact with the study participant. This individual will be informed that the research team is conducting a broad study on the relationship between individual and household health. Household interviews will chiefly comprise a subset of the battery administered to participants: specifically, the PHQ-9, WHODAS, and EQ-5D-3L (primary outcomes). In addition, household members will complete the BAS, as described above.

Process Evaluation. In the final year of the project, the investigators will conduct qualitative interviews to assess provider and patient experiences on their perceived effects of the intervention, as well as implementation barriers and strategies used to solve them. The goal is to identify key lessons learned, and to ready the intervention tools for scale-up at end of study.

Provider experience: In Year 5, the investigators will interview 10 clinical officers who prescribed ADT, as well as psychosocial counsellors who led PM+ sessions as well as diagnosed patients. In addition to discussing perceived strengths and weakness of the intervention and its implementation, the investigators will also discuss the training and supervision process, as well as provider job satisfaction and burnout.

Patient experience: A random sample of 20 participants (10 male, 10 female) will be interviewed after their final study assessment to assess their experiences with the intervention - including logistical aspect of participation, impact on personal mental health and wellbeing, as well as changes in relationships at the household level.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at integrated chronic care centers (IC3) in Neno District, Malawi
* Adult, age 18 or older

Exclusion Criteria:

* Psychosis, or indication of other Axis I psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms, 3 months | 3 months
  Depression symptoms will be measured with the Patient Health Questionnaire 9 (PHQ-9). This will be quantified as change in PHQ-9 score from baseline (pre-intervention) to 3-months (post-intervention).
Depression symptoms, 6 months | 6 months
  Depression symptoms will be measured with the Patient Health Questionnaire 9 (PHQ-9). This will be quantified as change in PHQ-9 score from baseline (pre-intervention) to 6-months (post-intervention).
Depression symptoms, 9 months | 9 months
  Depression symptoms will be measured with the Patient Health Questionnaire 9 (PHQ-9). This will be quantified as change in PHQ-9 score from baseline (pre-intervention) to 9-months (post-intervention).
Depression symptoms, 12 months | 12 months
  Depression symptoms will be measured with the Patient Health Questionnaire 9 (PHQ-9). This will be quantified as change in PHQ-9 score from baseline (pre-intervention) to 12-months (post-intervention).
Functional impairment, 3 months | 3 months
  Functional impairment will be measured with the World Health Organization (WHO) Disability Assessment Schedule (WHODAS). This will be quantified as change in WHODAS score from baseline (pre-intervention) to 3-months (post-intervention).
Functional impairment, 6 months | 6 months
  Functional impairment will be measured with the World Health Organization (WHO) Disability Assessment Schedule (WHODAS). This will be quantified as change in WHODAS score from baseline (pre-intervention) to 6-months (post-intervention).
Functional impairment, 9 months | 9 months
  Functional impairment will be measured with the World Health Organization (WHO) Disability Assessment Schedule (WHODAS). This will be quantified as change in WHODAS score from baseline (pre-intervention) to 9-months (post-intervention).
Functional impairment, 12 months | 12 months
  Functional impairment will be measured with the World Health Organization (WHO) Disability Assessment Schedule (WHODAS). This will be quantified as change in WHODAS score from baseline (pre-intervention) to 12-months (post-intervention).
Overall health profile, 3 months | 3 months
  A health profile will be generated for each individual using the EuroQol (EQ-5D-5L). This will be quantified as change in EQ-5D-5L score from baseline (pre-intervention) to 3-months (post-intervention).
Overall health profile, 6 months | 6 months
  A health profile will be generated for each individual using the EuroQol (EQ-5D-5L). This will be quantified as change in EQ-5D-5L score from baseline (pre-intervention) to 6-months (post-intervention).
Overall health profile, 9 months | 9 months
  A health profile will be generated for each individual using the EuroQol (EQ-5D-5L). This will be quantified as change in EQ-5D-5L score from baseline (pre-intervention) to 9-months (post-intervention).
Overall health profile, 12 months | 12 months
  A health profile will be generated for each individual using the EuroQol (EQ-5D-5L). This will be quantified as change in EQ-5D-5L score from baseline (pre-intervention) to 12-months (post-intervention).
Depression prevalence, 3 months | 3 months
  Depression prevalence will be quantified as the change in proportion of individuals with moderate-to-severe depression (PHQ-9>9) at each clinic from baseline (pre-intervention) to 3-months (post-intervention).
Depression prevalence, 6 months | 6 months
  Depression prevalence will be quantified as the change in proportion of individuals with moderate-to-severe depression (PHQ-9>9) at each clinic from baseline (pre-intervention) to 6-months (post-intervention).
Depression prevalence, 9 months | 9 months
  Depression prevalence will be quantified as the change in proportion of individuals with moderate-to-severe depression (PHQ-9>9) at each clinic from baseline (pre-intervention) to 9-months (post-intervention).
Depression prevalence, 12 months | 12 months
  Depression prevalence will be quantified as the change in proportion of individuals with moderate-to-severe depression (PHQ-9>9) at each clinic from baseline (pre-intervention) to 12-months (post-intervention).

SECONDARY OUTCOMES:
ART Adherence, 3 months | 3 months
  Among patients with HIV, ART adherence will be measured in terms of whether HIV+ enrollees have returned to an IC3 for antiretrovirals (ARVs) within the past three months. This will be quantified as change in adherence rates from baseline (pre-intervention) to 3-months (post-intervention)
ART Adherence, 6 months | 6 months
  Among patients with HIV, ART adherence will be measured in terms of whether HIV+ enrollees have returned to an IC3 for antiretrovirals (ARVs) within the past three months. This will be quantified as change in adherence rates from baseline (pre-intervention) to 6-months (post-intervention)
ART Adherence, 9 months | 9 months
  Among patients with HIV, ART adherence will be measured in terms of whether HIV+ enrollees have returned to an IC3 for antiretrovirals (ARVs) within the past three months. This will be quantified as change in adherence rates from baseline (pre-intervention) to 9-months (post-intervention)
ART Adherence, 12 months | 12 months
  Among patients with HIV, ART adherence will be measured in terms of whether HIV+ enrollees have returned to an IC3 for antiretrovirals (ARVs) within the past three months. This will be quantified as change in adherence rates from baseline (pre-intervention) to 12-months (post-intervention)
Viral suppression among HIV+ patients, 3 months | 3 months
  Viral load will be measured among patients with HIV (copies per milliliter). The investigators will examine change in the proportion of HIV+ patients who are virally-suppressed from baseline (pre-intervention) to 3-months (post-intervention)
Viral suppression among HIV+ patients, 6 months | 6 months
  Viral load will be measured among patients with HIV (copies per milliliter). The investigators will examine change in the proportion of HIV+ patients who are virally-suppressed from baseline (pre-intervention) to 6-months (post-intervention)
Viral suppression among HIV+ patients, 9 months | 9 months
  Viral load will be measured among patients with HIV (copies per milliliter). The investigators will examine change in the proportion of HIV+ patients who are virally-suppressed from baseline (pre-intervention) to 9-months (post-intervention)
Viral suppression among HIV+ patients, 12 months | 12 months
  Viral load will be measured among patients with HIV (copies per milliliter). The investigators will examine change in the proportion of HIV+ patients who are virally-suppressed from baseline (pre-intervention) to 12-months (post-intervention)
HIV disease staging among HIV+ patients, 3 months | 3 months
  Among HIV+, staging will be assessed according to WHO criteria. The investigators will examine change in the proportion of HIV+ patients with advanced disease staging from baseline (pre-intervention) to 3-months (post-intervention)
HIV disease staging among HIV+ patients, 6 months | 6 months
  Among HIV+, staging will be assessed according to WHO criteria. The investigators will examine change in the proportion of HIV+ patients with advanced disease staging from baseline (pre-intervention) to 6-months (post-intervention)
HIV disease staging among HIV+ patients, 9 months | 9 months
  Among HIV+, staging will be assessed according to WHO criteria. The investigators will examine change in the proportion of HIV+ patients with advanced disease staging from baseline (pre-intervention) to 9-months (post-intervention)
HIV disease staging among HIV+ patients, 12 months | 12 months
  Among HIV+, staging will be assessed according to WHO criteria. The investigators will examine change in the proportion of HIV+ patients with advanced disease staging from baseline (pre-intervention) to 12-months (post-intervention)
Systolic blood pressure among hypertensive patients, 3 months | 3 months
  Among patients with hypertension, systolic blood pressure (SBP) will be measured at routine clinic visits. The investigators will examine change in the proportion of hypertensive patients with SBP below 140 (over 90) from baseline (pre-intervention) to 3-months (post-intervention)
Systolic blood pressure among hypertensive patients, 6 months | 6 months
  Among patients with hypertension, systolic blood pressure (SBP) will be measured at routine clinic visits. The investigators will examine change in the proportion of hypertensive patients with SBP below 140 (over 90) from baseline (pre-intervention) to 6-months (post-intervention)
Systolic blood pressure among hypertensive patients, 9 months | 9 months
  Among patients with hypertension, systolic blood pressure (SBP) will be measured at routine clinic visits. The investigators will examine change in the proportion of hypertensive patients with SBP below 140 (over 90) from baseline (pre-intervention) to 9-months (post-intervention)
Systolic blood pressure among hypertensive patients, 12 months | 12 months
  Among patients with hypertension, systolic blood pressure (SBP) will be measured at routine clinic visits. The investigators will examine change in the proportion of hypertensive patients with SBP below 140 (over 90) from baseline (pre-intervention) to 12-months (post-intervention)
A1C levels among diabetic patients, 3 months | 3 months
  Among patients with diabetes, A1C (or random blood sugar) levels will be assessed at routine clinic visits. The investigators will examine change in the proportion of diabetic patients with controlled A1C / blood sugar levels from baseline (pre-intervention) to 3-months (post-intervention)
A1C levels among diabetic patients, 6 months | 6 months
  Among patients with diabetes, A1C (or random blood sugar) levels will be assessed at routine clinic visits. The investigators will examine change in the proportion of diabetic patients with controlled A1C / blood sugar levels from baseline (pre-intervention) to 6-months (post-intervention)
A1C levels among diabetic patients, 9 months | 9 months
  Among patients with diabetes, A1C (or random blood sugar) levels will be assessed at routine clinic visits. The investigators will examine change in the proportion of diabetic patients with controlled A1C / blood sugar levels from baseline (pre-intervention) to 9-months (post-intervention)
A1C levels among diabetic patients, 12 months | 12 months
  Among patients with diabetes, A1C (or random blood sugar) levels will be assessed at routine clinic visits. The investigators will examine change in the proportion of diabetic patients with controlled A1C / blood sugar levels from baseline (pre-intervention) to 12-months (post-intervention)
Number of seizures among patients with epilepsy, 3 months | 3 months
  Among patients with epilepsy, number of seizures will be documented during routine clinic visits. The investigator will examine change in the rate of seizures among epilepsy patients from baseline (pre-intervention) to 3-months (post-intervention)
Number of seizures among patients with epilepsy, 6 months | 6 months
  Among patients with epilepsy, number of seizures will be documented during routine clinic visits. The investigator will examine change in the rate of seizures among epilepsy patients from baseline (pre-intervention) to 6-months (post-intervention)
Number of seizures among patients with epilepsy, 9 months | 9 months
  Among patients with epilepsy, number of seizures will be documented during routine clinic visits. The investigator will examine change in the rate of seizures among epilepsy patients from baseline (pre-intervention) to 9-months (post-intervention)
Number of seizures among patients with epilepsy, 12 months | 12 months
  Among patients with epilepsy, number of seizures will be documented during routine clinic visits. The investigator will examine change in the rate of seizures among epilepsy patients from baseline (pre-intervention) to 12-months (post-intervention)

OTHER OUTCOMES:
Household member: burden of care | Pre-treatment (baseline) and 6-month follow-up
  Household burden of care will be evaluated with household members using a locally-adapted version of the Burden Assessment Schedule (BAS). This uses a 4 point ordinal scale from "not-at-all" (1) "to a lot" (4) and comprises 19-items, as detailed in Reinhard et al, 1994. A higher score indicates more significant (worse) burden of care. Investigators will examine change in continuous score on this measure.
Household member: depression | Pre-treatment (baseline) and 6-month follow-up
  Depression symptoms will be measured among household members using the Patient Health Questionnaire 9 (PHQ-9). This will be quantified as change in PHQ-9 score from baseline (pre-intervention) to 6-months (post-intervention).
Household member: functional impairment | Pre-treatment (baseline) and 6-month follow-up
  Functional impairment will be measured with the World Health Organization (WHO) Disability Assessment Schedule (WHODAS). This will be quantified as change in WHODAS score from baseline (pre-intervention) to 6-months (post-intervention).
Household member: overall health profile | Pre-treatment (baseline) and 6-month follow-up
  A health profile will be generated for each individual using the EuroQol (EQ-5D-5L). This will be quantified as change in EQ-5D-5L score from baseline (pre-intervention) to 3-months (post-intervention).
Perceived social support, 3 months | 3 months
  Patients will be assessed with the Multidimensional Scale of Perceived Social Support (MSPSS). This is a 12-item scale, with a 7-point ordinal scale from "very strongly disagree" (1) to "very strongly agree" (7), from Zimet et al. A higher score indicates greater (better) social support. This will be quantified as change in MSPSS from baseline to 3-months.
Perceived social support, 6 months | 6 months
  Patients will be assessed with the Multidimensional Scale of Perceived Social Support (MSPSS). This is a 12-item scale, with a 7-point ordinal scale from "very strongly disagree" (1) to "very strongly agree" (7), from Zimet et al. This will be quantified as change in MSPSS from baseline to 6-months.
Perceived social support, 9 months | 9 months
  Patients will be assessed with the Multidimensional Scale of Perceived Social Support (MSPSS). This is a 12-item scale, with a 7-point ordinal scale from "very strongly disagree" (1) to "very strongly agree" (7), from Zimet et al. This will be quantified as change in MSPSS from baseline to 9-months.
Perceived social support, 12 months | 12 months
  Patients will be assessed with the Multidimensional Scale of Perceived Social Support (MSPSS). This is a 12-item scale, with a 7-point ordinal scale from "very strongly disagree" (1) to "very strongly agree" (7), from Zimet et al. This will be quantified as change in MSPSS from baseline to 12-months.
Internalized mental health stigma, 3 months | 3 months
  Patients will be assessed with the Internalized Stigma of Mental Illness (ISMI-10) Scale, 1 10-item scale with a four-point ordinal scale from "strongly disagree (1) to "strongly agree" (4), developed by Boyd et al, 2014. A higher score indicates more (worse) stigma. This will be quantified as change in ISMI-10 from baseline (pre-intervention) to 3-months.
Internalized mental health stigma, 6 months | 6 months
  Patients will be assessed with the Internalized Stigma of Mental Illness (ISMI-10) Scale, 1 10-item scale with a four-point ordinal scale from "strongly disagree (1) to "strongly agree" (4), developed by Boyd et al, 2014. This will be quantified as change in ISMI-10 from baseline (pre-intervention) to 6-months.
Internalized mental health stigma, 9 months | 9 months
  Patients will be assessed with the Internalized Stigma of Mental Illness (ISMI-10) Scale, 1 10-item scale with a four-point ordinal scale from "strongly disagree (1) to "strongly agree" (4), developed by Boyd et al, 2014. This will be quantified as change in ISMI-10 from baseline (pre-intervention) to 9-months.
Internalized mental health stigma, 12 months | 12 months
  Patients will be assessed with the Internalized Stigma of Mental Illness (ISMI-10) Scale, 1 10-item scale with a four-point ordinal scale from "strongly disagree (1) to "strongly agree" (4), developed by Boyd et al, 2014. This will be quantified as change in ISMI-10 from baseline (pre-intervention) to 12-months.
AIDS-related stigma, 3 months | 3 months
  Patients with HIV will be assessed using the AIDS-Related Stigma Scale (ARSS), a 6-item scale using "disagree" vs. "agree" response options. A higher score indicates more (worse) stigma. This will be quantified as change in ARSS score from baseline (pre-intervention) to 3-months.
AIDS-related stigma, 6 months | 6 months
  Patients with HIV will be assessed using the AIDS-Related Stigma Scale (ARSS), a 6-item scale using "disagree" vs. "agree" response options. This will be quantified as change in ARSS score from baseline (pre-intervention) to 6-months.
AIDS-related stigma, 9 months | 9 months
  Patients with HIV will be assessed using the AIDS-Related Stigma Scale (ARSS), a 6-item scale using "disagree" vs. "agree" response options. This will be quantified as change in ARSS score from baseline (pre-intervention) to 9-months.
AIDS-related stigma, 12 months | 12 months
  Patients with HIV will be assessed using the AIDS-Related Stigma Scale (ARSS), a 6-item scale using "disagree" vs. "agree" response options. This will be quantified as change in ARSS score from baseline (pre-intervention) to 12-months.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners In Health, Neno, Neno District, Malawi

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, a data dictionary, and accompanying analytic code will be made available on Harvard University's DataVerse at the conclusion of the trial. Participants will be made aware of this during the informed consent process and provide their consent.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will become available in July 2025 and remain available at Harvard's DataVerse indefinitely.
Access Criteria: Access to data files on Harvard's DataVerse requires that researchers complete compliance and authorization forms.
URL: https://dataverse.harvard.edu/

REFERENCES:
- [Background] Udedi M. The prevalence of depression among patients and its detection by primary health care workers at Matawale Health Centre (Zomba). Malawi Med J. 2014 Jun;26(2):34-7. PMID 25157314
- [Background] World Economic Forum. The Global Economic Burden of Non-Communicable Diseases. World Economic Forum; Harvard School of Public Health; 2011.
- [Background] Passchier RV, Abas MA, Ebuenyi ID, Pariante CM. Effectiveness of depression interventions for people living with HIV in Sub-Saharan Africa: A systematic review & meta-analysis of psychological & immunological outcomes. Brain Behav Immun. 2018 Oct;73:261-273. doi: 10.1016/j.bbi.2018.05.010. Epub 2018 May 13. PMID 29768184
- [Background] McBain RK, Salhi C, Hann K, Kellie J, Kamara A, Salomon JA, Kim JJ, Betancourt TS. Improving outcomes for caregivers through treatment of young people affected by war: a randomized controlled trial in Sierra Leone. Bull World Health Organ. 2015 Dec 1;93(12):834-41. doi: 10.2471/BLT.14.139105. Epub 2015 Oct 16. PMID 26668435
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Mwale O, Mpinga K, Rukundo T, Kamwiyo M, Kayira W, Matanje B, Munyaneza F, Ruderman T, Raviola G, Smith S, Okunogbe A, Kachimanga C, McBain RK. Cost analysis of integrating depression treatment into chronic care in Malawi: evidence from a cluster randomised controlled trial. BMJ Open. 2025 Oct 7;15(10):e095494. doi: 10.1136/bmjopen-2024-095494. PMID 41062145
- [Derived] Mwale O, Kasambala C, Houde A, Mpinga K, Kayira W, Harawa M, Kamwiyo M, Isaacs R, Nhlema B, Ruderman T, Liwimbi O, Udedi M, Kelly K, McBain RK. Patient perspectives on group problem management plus for adults with major depressive disorder in rural Malawi. Glob Health Action. 2025 Dec;18(1):2500785. doi: 10.1080/16549716.2025.2500785. Epub 2025 May 9. PMID 40340587
- [Derived] McBain RK, Mwale O, Mpinga K, Kamwiyo M, Kayira W, Ruderman T, Connolly E, Watson SI, Wroe EB, Munyaneza F, Dullie L, Raviola G, Smith SL, Kulisewa K, Udedi M, Patel V, Wagner GJ. Effectiveness, cost-effectiveness, and positive externalities of integrated chronic care for adults with major depressive disorder in Malawi (IC3D): a stepped-wedge, cluster-randomised, controlled trial. Lancet. 2024 Nov 9;404(10465):1823-1834. doi: 10.1016/S0140-6736(24)01809-9. Epub 2024 Oct 30. PMID 39488229
- [Derived] Mpinga K, Rukundo T, Mwale O, Kamwiyo M, Thengo L, Ruderman T, Matanje B, Munyaneza F, Connolly E, Kulisewa K, Udedi M, Kachimanga C, Dullie L, McBain R. Depressive disorder at the household level: prevalence and correlates of depressive symptoms among household members. Glob Health Action. 2023 Dec 31;16(1):2241808. doi: 10.1080/16549716.2023.2241808. PMID 37554074
- [Derived] Mpinga K, Lee SD, Mwale O, Kamwiyo M, Nyirongo R, Ruderman T, Connolly E, Kayira W, Munyaneza F, Matanje B, Kachimanga C, Zaniku HR, Kulisewa K, Udedi M, Wagner G, McBain R. Prevalence and correlates of internalized stigma among adults with HIV and major depressive disorder in rural Malawi. AIDS Care. 2023 Nov;35(11):1775-1785. doi: 10.1080/09540121.2023.2195609. Epub 2023 Mar 31. PMID 37001058
- [Derived] McBain RK, Mwale O, Ruderman T, Kayira W, Connolly E, Chalamanda M, Kachimanga C, Khongo BD, Wilson J, Wroe E, Raviola G, Smith S, Coleman S, Kelly K, Houde A, Tebeka MG, Watson S, Kulisewa K, Udedi M, Wagner G. Stepped care for depression at integrated chronic care centers (IC3) in Malawi: study protocol for a stepped-wedge cluster randomized controlled trial. Trials. 2021 Sep 16;22(1):630. doi: 10.1186/s13063-021-05601-1. PMID 34530894

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT04777006/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT04777006/SAP_004.pdf